CLINICAL TRIAL: NCT05349864
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, 2-SEQUENCE, 3 PERIOD CROSSOVER STUDY TO EVALUATE THE EFFECT OF A LOW-FAT AND HIGH-FAT MEAL ON THE RELATIVE BIOAVAILABILITY OF PF-07284890 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Understand the Effect of Low-Fat and High-Fat Meals on the Medicine Called PF-07284890 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4471002
Record Dates: First submitted 2022-04-18; First posted 2022-04-27 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-08

CONDITIONS: Healthy Participants
Keywords: Food effect study

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07284890 Sequence 1 (Experimental): PF-07284890 tablet will be taken by mouth in a single dose for Treatment A while fasting.
  Five days later PF-07284890 tablet will be taken by mouth for Treatment B after a low fat meal.
  Five days later PF-07284890 tablet will be taken by mouth for Treatment C after a high fat meal.
  Interventions: Drug: PF-07284890 Treatment A; Drug: PF-07284890 Treatment B; Drug: PF-07284890 Treatment C
- PF-07284890 Sequence 2 (Experimental): PF-07284890 tablet will be taken by mouth for Treatment B after a low fat meal.
  Five days later PF-07284890 tablet will be taken by mouth in a single dose for Treatment A while fasting.
  Five days later PF-07284890 tablet will be taken by mouth for Treatment C after a high fat meal.
  Interventions: Drug: PF-07284890 Treatment A; Drug: PF-07284890 Treatment B; Drug: PF-07284890 Treatment C

INTERVENTIONS:
Drug: PF-07284890 Treatment A — PF-07284890 tablet by mouth while fasting
Drug: PF-07284890 Treatment B — PF-07284890 tablet after low fat meal
Drug: PF-07284890 Treatment C — PF-07284890 tablet after high fat meal

SUMMARY:
The purpose of the study is to evaluate the effect of a low-fat and high-fat meal on the medicine called PF-07284890 following three single doses PF-07284890. The study will include male participants and female participants of non-childbearing potential who are healthy. Participants will be required to stay in the clinical research unit for 15 days and 14 nights.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential and males who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and 12-lead ECGs.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant uveitis, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), including any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4471002

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-07284890 200 mg Fasted=>PF-07284890 200 mg Low-fat Meal=>PF-07284890 200 mg High-fat Meal: Participants in Sequence 1 received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under fasted conditions (Treatment A) in Period 1, followed by a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under low-fat meal fed conditions (Treatment B) in Period 2 after 5 days, and followed by a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under high-fat meal fed conditions (Treatment C) in Period 3 after 5 days.
- PF-07284890 200 mg Low-fat Meal=>PF-07284890 200 mg Fasted=>PF-07284890 200 mg High-fat Meal: Participants in Sequence 2 received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under low-fat meal fed conditions (Treatment B) in Period 1, followed by a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under fasted conditions (Treatment A) in Period 2 after 5 days, and followed by a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under high-fat meal fed conditions (Treatment C) in Period 3 after 5 days.
Period: Period 1 (5 Days)
Arm/Group | PF-07284890 200 mg Fasted=>PF-07284890 200 mg Low-fat Meal=>PF-07284890 200 mg High-fat Meal | PF-07284890 200 mg Low-fat Meal=>PF-07284890 200 mg Fasted=>PF-07284890 200 mg High-fat Meal
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2 (5 Days)
Arm/Group | PF-07284890 200 mg Fasted=>PF-07284890 200 mg Low-fat Meal=>PF-07284890 200 mg High-fat Meal | PF-07284890 200 mg Low-fat Meal=>PF-07284890 200 mg Fasted=>PF-07284890 200 mg High-fat Meal
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Period 3 (5 Days)
Arm/Group | PF-07284890 200 mg Fasted=>PF-07284890 200 mg Low-fat Meal=>PF-07284890 200 mg High-fat Meal | PF-07284890 200 mg Low-fat Meal=>PF-07284890 200 mg Fasted=>PF-07284890 200 mg High-fat Meal
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants assigned to the study intervention.
Groups:
- Female: The Female participant was a healthy adult of non-childbearing potential between 18-65 years of age.
- Male: Male participants were healthy adults between 18-65 years of age.
- Total: Total of all reporting groups
Arm/Group | Female | Male | Total
Number analyzed (Participants) | 1 | 11 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (NA) — Standard Deviation was not estimable due to insufficient number of participants with results. | 42.5 (12.23) | 43.8 (12.38)
Age, Customized [Count of Participants; unit: Participants]
  18-25 | 0 | 1 | 1
  26-35 | 0 | 1 | 1
  36-45 | 0 | 6 | 6
  >45 | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 11 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 10 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 4 | 4
  Black or African American | 1 | 5 | 6
  Asian | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PF-07284890 in Plasma, Comparison of Low-Fat Meal With Fasted Condition
Description: AUClast was defined as area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast). AUClast was determined by linear/Log trapezoidal method.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1 and 2
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest could be reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour per Milliliter (ng*hr/mL)
Groups:
- PF-07284890 200 mg Low-fat Meal (Test): Participants received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under low-fat meal fed conditions as the test treatment (Treatment B) in either Period 1 or Period 2.
- PF-07284890 200 mg Fasted (Reference): Participants received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under fasted conditions as the reference treatment (Treatment A) in either Period 1 or Period 2.
Arm/Group | PF-07284890 200 mg Low-fat Meal (Test) | PF-07284890 200 mg Fasted (Reference)
Number analyzed (Participants) | 12 | 12
Nanogram*Hour per Milliliter (ng*hr/mL) | 28270 (25) | 23510 (38)
Statistical Analysis 1: Comparison: PF-07284890 200 mg Low-fat Meal (Test) vs PF-07284890 200 mg Fasted (Reference); Test type: Equivalence — Using data from Treatment A and Treatment B, natural log transformed AUClast was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model, and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios; ratio of adjusted geometric means = 120.25, 90% CI 2-sided [109.76 to 131.75]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of PF-07284890 in Plasma, Comparison of Low-Fat Meal With Fasted Condition
Description: AUCinf was defined as area under the plasma concentration-time curve from time zero extrapolated to infinity. AUCinf = AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1 and 2
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest could be reported. Overall number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07284890 200 mg Low-fat Meal (Test) | PF-07284890 200 mg Fasted (Reference)
Number analyzed (Participants) | 9 | 8
ng*hr/mL | 29380 (25) | 24600 (46)
Statistical Analysis 1: Comparison: PF-07284890 200 mg Low-fat Meal (Test) vs PF-07284890 200 mg Fasted (Reference); Test type: Equivalence — Using data from Treatment A and Treatment B, natural log transformed AUCinf was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model, and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios; ratio of adjusted geometric means = 116.22, 90% CI 2-sided [97.91 to 137.95]

3. Primary Outcome: Maximum Observed Concentration (Cmax) of PF-07284890 in Plasma, Comparison of Low-Fat Meal With Fasted Condition
Description: Cmax was defined as maximum observed plasma concentration. The determination method of Cmax was observing directly from data.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1 and 2
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 concentration value could be reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | PF-07284890 200 mg Low-fat Meal (Test) | PF-07284890 200 mg Fasted (Reference)
Number analyzed (Participants) | 12 | 12
Nanogram per Milliliter (ng/mL) | 3460 (19) | 1672 (43)
Statistical Analysis 1: Comparison: PF-07284890 200 mg Low-fat Meal (Test) vs PF-07284890 200 mg Fasted (Reference); Test type: Equivalence — Using data from Treatment A and Treatment B, natural log transformed Cmax was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model, and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios; ratio of adjusted geometric means = 206.91, 90% CI 2-sided [171.14 to 250.15]

4. Primary Outcome: AUClast of PF-07284890 in Plasma, Comparison of High-Fat Meal With Fasted Condition
Description: as for outcome 1
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1-3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- PF-07284890 200 mg High-fat Meal (Test): Participants received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under high-fat meal fed conditions as the test treatment (Treatment C) in Period 3.
Arm/Group | PF-07284890 200 mg High-fat Meal (Test) | PF-07284890 200 mg Fasted (Reference)
Number analyzed (Participants) | 10 | 12
ng*hr/mL | 31300 (21) | 23510 (38)
Statistical Analysis 1: Comparison: PF-07284890 200 mg High-fat Meal (Test) vs PF-07284890 200 mg Fasted (Reference); Test type: Equivalence — Using data from Treatment A and Treatment C, natural log transformed AUClast was analyzed using a mixed effect model with treatment and sequence as a fixed effect and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model, and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios; ratio of adjusted geometric means = 135.77, 90% CI 2-sided [114.36 to 161.19]

5. Primary Outcome: AUCinf of PF-07284890 in Plasma, Comparison of High-Fat Meal With Fasted Condition
Description: as for outcome 2
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1-3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07284890 200 mg High-fat Meal (Test) | PF-07284890 200 mg Fasted (Reference)
Number analyzed (Participants) | 7 | 8
ng*hr/mL | 34130 (20) | 24600 (46)
Statistical Analysis 1: Comparison: PF-07284890 200 mg High-fat Meal (Test) vs PF-07284890 200 mg Fasted (Reference); Test type: Equivalence — Using data from Treatment A and Treatment C, natural log transformed AUCinf was analyzed using a mixed effect model with treatment and sequence as a fixed effect and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model, and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios; ratio of adjusted geometric means = 138.36, 90% CI 2-sided [106.11 to 180.41]

6. Primary Outcome: Cmax of PF-07284890 in Plasma, Comparison of High-Fat Meal With Fasted Condition
Description: as for outcome 3
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1-3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07284890 200 mg High-fat Meal (Test) | PF-07284890 200 mg Fasted (Reference)
Number analyzed (Participants) | 10 | 12
ng/mL | 3892 (22) | 1672 (43)
Statistical Analysis 1: Comparison: PF-07284890 200 mg High-fat Meal (Test) vs PF-07284890 200 mg Fasted (Reference); Test type: Equivalence — Using data from Treatment A and Treatment C, natural log transformed Cmax was analyzed using a mixed effect model with treatment and sequence as a fixed effect and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model, and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios; ratio of adjusted geometric means = 236.58, 90% CI 2-sided [190.12 to 294.38]

7. Secondary Outcome: Time to Reach Cmax (Tmax) of PF-07284890 in Plasma
Description: Tmax was defined as time to reach maximum observed plasma concentration. The determination method of Tmax was observing directly from data as time of first occurrence.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1-3
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours (hr)
Groups:
- PF-07284890 200 mg Fasted: Participants received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under fasted conditions (Treatment A) in either Period 1 or Period 2.
- PF-07284890 200 mg Low-fat Meal: Participants received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under low-fat meal fed conditions (Treatment B) in either Period 1 or Period 2.
- PF-07284890 200 mg High-fat Meal: Participants received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under high-fat meal fed conditions (Treatment C) in Period 3.
Arm/Group | PF-07284890 200 mg Fasted | PF-07284890 200 mg Low-fat Meal | PF-07284890 200 mg High-fat Meal
Number analyzed (Participants) | 12 | 12 | 10
Hours (hr) | 3.00 [1.00 to 4.00] | 3.00 [2.00 to 4.02] | 4.01 [2.00 to 8.00]

8. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of PF-07284890 in Plasma
Description: t1/2 was defined as the time required for the plasma concentration to decline by 50% during the elimination phase. t1/2 = loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1-3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-07284890 200 mg Fasted | PF-07284890 200 mg Low-fat Meal | PF-07284890 200 mg High-fat Meal
Number analyzed (Participants) | 8 | 9 | 7
hr | 16.36 (4.1925) | 17.73 (5.2538) | 16.19 (4.4712)

9. Secondary Outcome: Apparent Clearance (CL/F) of PF-07284890 in Plasma
Description: CL/F was defined as the apparent clearance. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). CL/F = dose/AUCinf, where AUCinf was the area under the plasma concentration-time curve from time zero extrapolated to infinity.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1-3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per Hour (L/hr)
Arm/Group | PF-07284890 200 mg Fasted | PF-07284890 200 mg Low-fat Meal | PF-07284890 200 mg High-fat Meal
Number analyzed (Participants) | 8 | 9 | 7
Liter per Hour (L/hr) | 8.130 (46) | 6.810 (25) | 5.860 (20)

10. Secondary Outcome: Apparent Volume of Distribution for Extravascular Dosing (Vz/F) of PF-07284890 in Plasma
Description: Vz/F was defined as the apparent volume of distribution for extravascular dosing. Determination method of Vz/F was dose/(AUCinf*kel), where kel was the terminal phase rate constant calculated by a linear regression of the loglinear concentration-time curve.
Time Frame: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose of PF-07284890 in Periods 1-3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | PF-07284890 200 mg Fasted | PF-07284890 200 mg Low-fat Meal | PF-07284890 200 mg High-fat Meal
Number analyzed (Participants) | 8 | 9 | 7
Liter (L) | 186.4 (36) | 168.5 (30) | 132.9 (12)

11. Secondary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Any events occurring following start of treatment were considered as TEAEs.
Time Frame: From baseline up to 35 days after last dose of PF-07284890, up to 11 weeks
Population: The analysis population included all participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07284890 200 mg Fasted | PF-07284890 200 mg Low-fat Meal | PF-07284890 200 mg High-fat Meal
Number analyzed (Participants) | 12 | 12 | 10
Participants | 5 | 3 | 2

12. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: The hematological (Lymphocytes/Leukocytes, Neutrophils/Leukocytes and Monocytes/Leukocytes), clinical chemistry (Urate and Potassium) and urinalysis (Urine Hemoglobin, Leukocyte Esterase and Bacteria) safety tests were assessed against the pre-specified criteria. The assessment did not take into account whether each participant's baseline test result was within or outside the laboratory reference range for the particular laboratory parameter.
Time Frame: From baseline up to 35 days after last dose of PF-07284890, up to 11 weeks
Population: The analysis population included all participants assigned to study intervention and who took at least 1 dose of study intervention. Number of Participants Analyzed = number of participants evaluable for laboratory abnormalities. Number Analyzed = total number of participants with at least one observation of the given laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07284890 200 mg Fasted | PF-07284890 200 mg Low-fat Meal | PF-07284890 200 mg High-fat Meal
Number analyzed (Participants) | 12 | 12 | 10
Participants
  Lymphocytes/Leukocytes >1.2 x upper limit of normal (ULN) | 0 | 0 | 1
  Neutrophils/Leukocytes <0.8 x lower limit of normal (LLN) | 0 | 0 | 1
  Monocytes/Leukocytes >1.2 x ULN | 1 | 1 | 1
  Urate >1.2 x ULN | 0 | 1 | 0
  Potassium >1.1 x ULN | 0 | 1 | 0
  Urine Hemoglobin >=1 | 0 | 1 | 0
  Leukocyte Esterase >=1 | 0 | 0 | 1
  Bacteria >20: number analyzed (Participants) | 0 | 1 | 1
  Bacteria >20 | 0 | 1 | 0

13. Secondary Outcome: Number of Participants With Pre-Specified Categorization Criteria for Vital Signs
Description: Supine systolic/diastolic blood pressure (BP) and pulse rate (PR) were measured and evaluated against pre-specified categorization criteria. The criteria included change of supine systolic/diastolic BP >=30 mmHg increase or decrease, and value of supine PR >120 beats per minute (bpm).
Time Frame: From baseline up to 35 days after last dose of PF-07284890, up to 11 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07284890 200 mg Fasted | PF-07284890 200 mg Low-fat Meal | PF-07284890 200 mg High-fat Meal
Number analyzed (Participants) | 12 | 12 | 10
Participants
  Change of Supine Systolic BP >=30 mmHg Increase | 0 | 0 | 0
  Change of Supine Systolic BP >=30 mmHg Decrease | 0 | 0 | 0
  Change of Supine Diastolic BP >=20 mmHg Increase | 0 | 0 | 0
  Change of Supine Diastolic BP >=20 mmHg Decrease | 0 | 0 | 0
  Value of Supine PR >120 bpm | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Pre-Specified Categorization Criteria for 12-Lead Electrocardiograms (ECGs)
Description: Standard 12-lead ECGs utilizing limb leads were collected using an ECG machine that automatically calculated the heart rate (HR) and measured PR interval, QT interval, corrected QT interval using Fridericia's formula (QTcF), and time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS) complex. The number of participants with PR/QRS values and percent change from baseline, QT interval values, and QTcF values and increases from baseline in the pre-specified categories were summarized in this outcome measure (OM).
Time Frame: From baseline up to 35 days after last dose of PF-07284890, up to 11 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07284890 200 mg Fasted | PF-07284890 200 mg Low-fat Meal | PF-07284890 200 mg High-fat Meal
Number analyzed (Participants) | 12 | 12 | 10
Participants
  Value of PR Interval >=300 msec | 0 | 0 | 0
  Percent Change of PR Interval >=25/50% | 0 | 0 | 0
  Value of QRS Duration >=140 msec | 0 | 0 | 0
  Percent Change of QRS Duration >=50% | 0 | 0 | 0
  Value of QT Interval >=500 msec | 0 | 0 | 0
  Value of QTcF >450 msec and <=480 msec | 0 | 0 | 1
  Value of QTcF >480 msec and <=500 msec | 0 | 0 | 0
  Value of QTcF >500 msec | 0 | 0 | 0
  Change of QTcF >=30 msec and <=60 msec | 0 | 0 | 2
  Change of QTcF >60 msec | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline up to 35 days after last dose of PF-07284890, up to 11 weeks
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Groups:
- PF-07284890 200 mg Fasted in Period 1 (Sequence 1): Participants in Sequence 1 received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under fasted conditions (Treatment A) in Period 1.
- PF-07284890 200 mg Low-fat Meal in Period 1 (Sequence 2): Participants in Sequence 2 received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under low-fat meal fed conditions (Treatment B) in Period 1.
- PF-07284890 200 mg Low-fat Meal in Period 2 (Sequence 1): Participants in Sequence 1 received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under low-fat meal fed conditions (Treatment B) in Period 2.
- PF-07284890 200 mg Fasted in Period 2 (Sequence 2): Participants in Sequence 2 received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under fasted conditions (Treatment A) in Period 2.
- PF-07284890 200 mg High-fat Meal in Period 3 (Sequence 1): Participants in Sequence 1 received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under high-fat meal fed conditions (Treatment C) in Period 3.
- PF-07284890 200 mg High-fat Meal in Period 3 (Sequence 2): Participants in Sequence 2 received a single oral dose of PF-07284890 200 mg (2 × 100 mg tablets) under high-fat meal fed conditions (Treatment C) in Period 3.
Arm/Group | PF-07284890 200 mg Fasted in Period 1 (Sequence 1) | PF-07284890 200 mg Low-fat Meal in Period 1 (Sequence 2) | PF-07284890 200 mg Low-fat Meal in Period 2 (Sequence 1) | PF-07284890 200 mg Fasted in Period 2 (Sequence 2) | PF-07284890 200 mg High-fat Meal in Period 3 (Sequence 1) | PF-07284890 200 mg High-fat Meal in Period 3 (Sequence 2)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 2/6 | 3/6 | 1/5 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07284890 200 mg Fasted in Period 1 (Sequence 1) (N=6) | PF-07284890 200 mg Low-fat Meal in Period 1 (Sequence 2) (N=6) | PF-07284890 200 mg Low-fat Meal in Period 2 (Sequence 1) (N=6) | PF-07284890 200 mg Fasted in Period 2 (Sequence 2) (N=6) | PF-07284890 200 mg High-fat Meal in Period 3 (Sequence 1) (N=5) | PF-07284890 200 mg High-fat Meal in Period 3 (Sequence 2) (N=5)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT05349864/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT05349864/SAP_001.pdf